CLINICAL TRIAL: NCT03486808
Title: Effect of Dual Site-Dual Channel Non-invasive Brain Stimulation for Recovery of Language and Cognitive Function in Healthy Subjects
Brief Title: Dual Site-Dual Channel Non-invasive Brain Stimulation for Language and Cognitive Function in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-08-124-D
Record Dates: First submitted 2018-03-22; First posted 2018-04-03 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: transcranial direct current stimulation; motor function

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dual stimulation (Experimental): i) anodal stimulation of left inferior frontal cortex ii) anodal stimulation on left dorsolateral prefrontal cortex
  Interventions: Device: IFG stimulation; Device: DLPFC stimulation
- IFG stimulation (Active Comparator): anodal stimulation of left inferior frontal cortex
  Interventions: Device: IFG stimulation
- DLPFC stimulation (Active Comparator): anodal stimulation on left dorsolateral prefrontal cortex
  Interventions: Device: DLPFC stimulation
- Sham stimulation (Sham Comparator): sham stimulation
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: IFG stimulation — stimulating left inferior frontal cortex with transcranial direct current stimulation for 30 minutes
  Arms: Dual stimulation; IFG stimulation
Device: DLPFC stimulation — stimulating left dorsolateral prefrontal cortex with transcranial direct current stimulation for 30 minutes
  Arms: DLPFC stimulation; Dual stimulation
Device: Sham stimulation — sham stimulation over both left inferior frontal cortex and dorsolateral prefrontal cortex
  Arms: Sham stimulation

SUMMARY:
The aim of this study is to investigate the effect of dual site-dual channel non-invasive brain stimulation for recovery of language and cognitive function in healthy. Simultaneous dual site-dual channel stimulation was applied by using two sets of transcranial direct current stimulation devices. All subjects will go through four conditions of transcranial direct current stimulation with for 30 minutes. Four conditions are 1) Dual stimulation: i) anodal stimulation on left inferior frontal cortex, ii) anodal stimulation on left dorsolateral prefrontal cortex. 2) IFG stimulation: anodal stimulation on left inferior frontal cortex; 3) DLPFC stimulation: anodal stimulation on left dorsolateral prefrontal cortex area. 4) sham stimulation

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects with age over 19 years old

Exclusion Criteria:

* history of disorders involving central nervous system
* patients with severe medical or psychiatric disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Korean Boston naming test | Baseline and after intervention (approximately 30 minutes)
  measures naming ability thorough picture naming test
Verbal 3 back test | Baseline and after intervention (approximately 30 minutes)
  measure working memory

SECONDARY OUTCOMES:
Korean Color Word Stroop test | Baseline and after intervention (approximately 30 minutes)
  measures selective attention and executive function
Controlled Oral Word Association Test | Baseline and after intervention (approximately 30 minutes)
  measure verbal fluency

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided